CLINICAL TRIAL: NCT03462043
Title: A Pivotal, Open-Label, Randomized, Crossover Study in Patients With Advanced Parkinson's Disease to Assess the Relative Bioavailability of Levodopa Administered as ND0612 Subcutaneous Infusion Versus Levodopa Administered as Carbidopa-Levodopa Enteral Suspension
Brief Title: A Study in Patients With Advanced Parkinson's Disease to Assess the Relative Bioavailability of Levodopa Administered as ND0612 Subcutaneous Infusion Versus Levodopa Administered as Carbidopa-Levodopa Enteral Suspension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to change the study design
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ND0612-315
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Parkinson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Sequence A (Active Comparator)
  Interventions: Combination Product: ND0612; Combination Product: CLES
- Sequence B (Active Comparator)
  Interventions: Combination Product: ND0612; Combination Product: CLES
- Sequence C (Active Comparator)
  Interventions: Combination Product: ND0612; Combination Product: CLES
- Sequence D (Active Comparator)
  Interventions: Combination Product: ND0612; Combination Product: CLES

INTERVENTIONS:
Combination Product: ND0612 — s.c. infused
Combination Product: CLES — Carbidopa-Levodopa Enteral Suspension.

SUMMARY:
This study will assess the relative bioavailability of s.c. infused ND0612 versus jejunally infused CLES in patients with advanced PD.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, crossover study to assess the relative bioavailability of s.c. infused ND0612 versus jejunally infused CLES in patients with advanced PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Advanced PD treated with LD/CD at a dose of at least 800 mg LD
* Female patients must have a negative pregnancy test at screening and at admission.
* Patients must have a body mass index (BMI) within the range of 18.5 - 35 kg/m2, where BMI = body weight (kg) / height (m2) at screening.
* Must be willing and able to communicate and participate in the whole study.
* Must provide written informed consent.
* Must agree to use an adequate method of contraception (per local independent ethics committee requirements).
* Area of administration to be evaluable for local skin reaction (normal skin without skin burns, scars or large tattoos in the area of administration

Exclusion Criteria:

* Any relevant medical, surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the Investigator, makes the patient unsuitable for study entry or potentially unable to complete all aspects of the study.
* Positive serum serology for Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV) at the screening visit.
* Patients with a history of drug abuse or alcoholism within the past 12 months prior to screening or positive drugs of abuse or alcohol test result at the screening visit and/or on admission.
* Clinically significant electrocardiogram (ECG) rhythm abnormalities.
* Renal or liver dysfunction that may alter drug metabolism including: serum creatinine >1.5 mg/dL, serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 x upper limit of normal (ULN), total serum bilirubin >2.5 mg/dL.
* Psychiatric, neurological or behavioral disorders that may interfere with the conduct or interpretation of the study, including dementia, or patients who are considered to be violent or at suicidal risk by the Investigator.
* Blood loss of greater than 500 mL within the previous 3 months prior to first dosing.
* use of any medication from the prohibited concomitant therapies

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-11-20 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Bioavailability | 6-7 days
  To assess relative bioavailability of levodopa (LD) administered as ND0612, infused subcutaneously (s.c.), versus LD administered as carbidopa-levodopa enteral suspension (CLES)

CONTACTS AND LOCATIONS:
Overall Officials: Osnat Ehrman, Study Director — NeuroDerm Ltd.
Locations (1):
- 91601, Roma, Italy